CLINICAL TRIAL: NCT05814562
Title: Cardiovascular Precision Medicine & Remote Intervention - Pilot Protocol
Brief Title: Cardiovascular Precision Medicine & Remote Intervention
Acronym: CP&R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Edward-Elmhurst Health System (Other)
Responsible Party: Principal Investigator, Eyal Shemesh, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00680
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Pre-intervention versus post intervention evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote Intervention (Experimental): An automatic blood pressure monitor will be given to patients upon enrollment. During the three months after enrollment, patients will be administered remote intervention weekly during the first month, and biweekly during the second and third month. At the onset of those sessions the patients will be asked to measure their blood pressure and this will be recorded by the coordinator.
  Interventions: Behavioral: Remote Intervention

INTERVENTIONS:
Behavioral: Remote Intervention — The study utilizes a tailored telemetric intervention to improve adherence to medications. The telemetric intervention (administered via telephone, or interactive internet chat applications such as Zoom ©, FaceTime ® or Skype ®) will enable experienced therapists to address nonadherence from a remote location, using a structured, tailored approach that accommodates specific patient needs.

SUMMARY:
This exploratory / proof of concept study aims to evaluate whether it is possible to identify at-risk patients based on EHR review of blood pressure fluctuation over time and cholesterol levels, recruit those patients, and engage them in a remote intervention protocol.

DETAILED DESCRIPTION:
Patients will be screened for participation based on EHR blood pressure measurements. Those who potential meet the prespecified criteria will be approached during a clinic visits about participation in the study. Patients who agree to participate and sign an informed consent will be given an automatic blood pressure monitor and their contact details will be obtained in order to enable administration of the intervention.

The intervention's theoretical underpinnings are principles previously identified as promising or helpful in health care management of at-risk patients. The principles are:

1. "Hovering", using a risk marker, to guide an intervention
2. Addressing posttraumatic avoidance as a way to improve adherence, using an imaginal exposure paradigm.
3. Using a remote interventionist via a telemetric interface that involves active, dynamic patient engagement rather than automated processes

ELIGIBILITY:
Participants will be screened for eligibility using the eligibility criteria delineated below. Informed Consent will be obtained for eligible candidates.

Inclusion Criteria:

The patient must meet all of below criteria to be eligible for enrollment in the study:

* The patient is > 18 years of age at enrollment.
* The patient is followed at the cardiology clinic and was diagnosed with hypertension and hypercholesterolemia more than 12 months prior to EHR screening, and has been prescribed at least one antihypertensive medication and at least one lipid-lowering agent over the 6 months prior to EHR screening
* The patient can be reached either by phone or via an internet-enabled device.
* The patient speaks English or Spanish at a level that allows them to understand the study procedures and consent to the study.
* The coefficient of Variation (CoV) of at least three systolic blood pressure measurements present in the EHR over the 12 months prior to EHR screening is > 10%.

Exclusion Criteria:

None of the following may be present if the patient is to be eligible for enrollment in the study:

* The patient is suffering from a psychiatric or developmental disorder that prevents him or her from understanding the protocol or engaging in the intervention (e.g., autistic disorder, psychosis).
* The investigator determines that a remote intervention paradigm is not advisable because of specific patient or environmental characteristics (investigator discretion).
* The patient is suffering from a medical disorder that makes control of blood pressure especially challenging or unlikely (e.g., end stage renal disease, uncontrolled endocrine disorders)
* Unstable blood pressure or hyperlipidemia that may require change in therapy in the 3 months after enrolment
* Significant heart failure (NYHA > 2) or ejection fraction < 50%
* Recent thromboembolic events such as a myocardial infarction, stroke, acute coronary syndrome, transient ischemic attack in the 6 months prior to enrolment
* Any arrythmia requiring medical or device therapy within 6 months prior to enrolment.
* The patient is hospitalized or was hospitalized in the last 6 months prior to enrollment. Patients hospitalized after enrollment are not excluded.

PI decision to exclude (for example - PI determines that the patient may be harmed by the study for a reason that is not covered by the exclusion criteria)

Withdrawal Criteria

Participants will be withdrawn from the intervention if they wish to not be called anymore. If they agree to continue to have their data collected from the medical chart, they would not be withdrawn from the study. Patients will be withdrawn from the study (their pre-withdrawal data will be used for the primary intent-to-treat analysis unless prohibited) for the following reasons:

* The patient dies.
* The patient becomes psychotic as defined in DSM-V, or suffers from an event that makes him or her unable to participate in the intervention (e.g. loss of hearing, loss of cognitive ability).
* The patient's care is transferred to another center, and it is impossible to get the primary and secondary outcome data.
* Patient decision
* Investigator decision
* DSMC or IRB determination related to the occurrence of an adverse event, or for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Blood pressure readings | Baseline and Week 12
  The change in systolic blood pressure from Visit 1 (enrollment) to Visit 9 (week 12) will be tested using a paired t-test. Changes will be based on measures taken with the same monitor (clinic or home) at both time points if possible; if changes with both clinic and home monitors are available, then measures using the clinic monitor will be used.
  Blood pressure readings (min max mean and fluctuation) before the intervention commences and during and after it, in an intent-to treat paradigm.

SECONDARY OUTCOMES:
Change in Blood Pressure Variability Index | 6 months prior to screening and Week 2
  A blood pressure variability index (BPVI) will be defined as the standard deviation (SD) of selected blood pressure measurements. A BPCoV will also be defined as the coefficient of variation of selected systolic blood pressure measurements. The BPVI over the 6 months prior to EHR screening (at least 3 measurements per eligibility criteria); and of measures at study visit at week 2 will be computed. BPCoV measures will be computed analogously. If no measure is available at a particular week, the closest measure in time will be used. Only patients with at least 3 post-enrollment BP measurements will be included in the analyses. Measures before and after enrollment will be compared with a paired t-test. BPVI will be considered the primary analysis, with analysis of BPCoV supportive.
Change in Blood Pressure Variability Index | 6 months prior to screening and Week 4
  A blood pressure variability index (BPVI) will be defined as the standard deviation (SD) of selected blood pressure measurements. A BPCoV will also be defined as the coefficient of variation of selected systolic blood pressure measurements. The BPVI over the 6 months prior to EHR screening (at least 3 measurements per eligibility criteria); and of measures at study visit at week 4 will be computed. BPCoV measures will be computed analogously. If no measure is available at a particular week, the closest measure in time will be used. Only patients with at least 3 post-enrollment BP measurements will be included in the analyses. Measures before and after enrollment will be compared with a paired t-test. BPVI will be considered the primary analysis, with analysis of BPCoV supportive.
Change in Blood Pressure Variability Index | 6 months prior to screening and Week 8
  A blood pressure variability index (BPVI) will be defined as the standard deviation (SD) of selected blood pressure measurements. A BPCoV will also be defined as the coefficient of variation of selected systolic blood pressure measurements. The BPVI over the 6 months prior to EHR screening (at least 3 measurements per eligibility criteria); and of measures at study visit at week 8 will be computed. BPCoV measures will be computed analogously. If no measure is available at a particular week, the closest measure in time will be used. Only patients with at least 3 post-enrollment BP measurements will be included in the analyses. Measures before and after enrollment will be compared with a paired t-test. BPVI will be considered the primary analysis, with analysis of BPCoV supportive.
Change in Blood Pressure Variability Index | 6 months prior to screening and Week 12
  A blood pressure variability index (BPVI) will be defined as the standard deviation (SD) of selected blood pressure measurements. A BPCoV will also be defined as the coefficient of variation of selected systolic blood pressure measurements. The BPVI over the 6 months prior to EHR screening (at least 3 measurements per eligibility criteria); and of measures at study visit at 12 will be computed. BPCoV measures will be computed analogously. If no measure is available at a particular week, the closest measure in time will be used. Only patients with at least 3 post-enrollment BP measurements will be included in the analyses. Measures before and after enrollment will be compared with a paired t-test. BPVI will be considered the primary analysis, with analysis of BPCoV supportive.
Proportion of clinic patients "at risk" | Baseline
  The proportion of patients who display an "at risk" pattern will be computed as the number of patients with a CoV of at least three systolic blood pressure measurements present in the EHR over the 6 months prior to screening > 10% out of the number of patients meeting all eligibility criteria identifiable during screening of the EHR. The proportion and its associated 90% CI will be presented.
Proportion of high risk who agree to participate | Baseline
  The proportion of "high risk" patients who agree to participate will be computed as the number of patients who sign the informed consent form out of the number of patients identified as meeting all study eligibility criteria and approached for informed consent. The proportion and its associated 90% CI will be presented.
Proportion of high risk patients successfully engaged | 12 weeks
  The proportion of "high risk" patients successfully engaged will be computed as the number of patients who participate in 3 more more remote intervention sessions out of the number of patients who agree to participate in the study. The proportion and its associated 90% CI will be presented.
Change in cholesterol level | Visit 1 (Week 0) and Visit 9 (Week 12)
  The changes from in total, LDL, HDL cholesterol levels; and in triglyceride levels from Visit 1 (enrollment; defined as the last measure taken for clinical reasons prior to consent or during the visit in which consent was obtained) to Visit 9 (week 12) will be tested using paired t-tests.
Change in blood pressure | Visit 1 (Week 0) and Visit 9 (Week 12)
  The change in systolic blood pressure from Visit 1 (enrollment) to Visit 9 (week 12) will be tested using a paired t-test. Changes will be based on measures taken with the same monitor (clinic or home) at both time points if possible; if changes with both clinic and home monitors are available, then measures using the clinic monitor will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Deborah Reynolds, MD, Principal Investigator — Edward-Elmhurst Health System
Locations (1):
- Elmhurst Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study

REFERENCES:
- [Derived] Shemesh E, Reynolds D, Sidhu J, Duncan-Park S, Tejiram RA, Davison BA, Takagi K, Edwards C, Rubinstein D, Annunziato RA, Cotter G. Reducing blood pressure variability-results from a single-arm proof of concept prospective trial. Sci Rep. 2025 Aug 12;15(1):29449. doi: 10.1038/s41598-025-14968-z. PMID 40790229
- [Derived] Reynolds D, Annunziato RA, Sidhu J, Cotter G, Davison BA, Takagi K, Duncan-Park S, Rubinstein D, Shemesh E. Cardiovascular Precision Medicine and Remote Intervention Trial Rationale and Design. J Clin Med. 2024 Oct 21;13(20):6274. doi: 10.3390/jcm13206274. PMID 39458224